CLINICAL TRIAL: NCT03412890
Title: LIBERTY EXTENSION: An International Phase 3 Open-Label, Single-Arm, Long-Term Efficacy and Safety Extension Study to Evaluate Relugolix Co-Administered With Low-Dose Estradiol and Norethindrone Acetate in Women With Heavy Menstrual Bleeding Associated With Uterine Fibroids
Brief Title: LIBERTY EXTENSION: Efficacy and Safety Extension Study of Relugolix in Women With Heavy Menstrual Bleeding Associated With Uterine Fibroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Myovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVT-601-3003; 2017-003310-74 (EudraCT Number)
Record Dates: First submitted 2018-01-19; First posted 2018-01-29 (Actual); Results first posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Heavy Menstrual Bleeding; Uterine Fibroid
Keywords: Uterine Fibroid; Heavy Menstrual Bleeding; Menstrual Blood Volume
MeSH Terms: conditions — Menorrhagia; Leiomyoma | interventions — relugolix; estradiol, norethindrone drug combination

STUDY DESIGN:
Intervention Model Description: Open-Label Extension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Relugolix plus E2/NETA (Experimental): Relugolix co-administered with E2/NETA for 28 weeks.
  Interventions: Drug: Relugolix; Drug: Estradiol/norethindrone acetate

INTERVENTIONS:
Drug: Relugolix — Relugolix 40-mg tablet administered orally once daily
  Other Names: MVT-601; TAK-385
Drug: Estradiol/norethindrone acetate — Capsule containing co-formulated tablet of E2 (1 mg) and NETA (0.5 mg) administered orally once daily
  Other Names: E2/NETA

SUMMARY:
The purpose of this study was to determine the long-term efficacy and safety of relugolix 40 milligrams (mg) once daily co-administered with estradiol (E2) and norethindrone acetate (NETA) for 28 weeks on heavy menstrual bleeding associated with uterine fibroids in participants who previously completed a 24-week treatment period in one of the pivotal studies (MVT-601-3001 or MVT-601-3002).

DETAILED DESCRIPTION:
This study is an international phase 3 open-label, single-arm, long-term efficacy and safety extension study that enrolled eligible participants who have completed their participation in one of the phase 3 randomized, double-blind, placebo-controlled pivotal studies, MVT-601-3001 (LIBERTY 1 - NCT03049735) or MVT-601-3002 (LIBERTY 2 - NCT 03103087). All participants received relugolix 40 mg orally once daily co-administered with E2 (1 mg) and NETA (0.5 mg) for 28 weeks.

Approximately 600 women with heavy menstrual bleeding associated with uterine fibroids were to be enrolled, after having completed a 24-week treatment period in one of the pivotal studies. The objectives of the study were to evaluate long-term efficacy and safety through up to 52 weeks of treatment (including treatment during the pivotal study) of relugolix co-administered with E2/NETA.

Screening and baseline procedures were to be done at the same visit for this extension study (referred to as the "Week 24/Baseline Visit"), which coincided with the Week 24 Visit from the pivotal study and was to be defined as the date of completion of the last Week 24 procedure in the pivotal study. Participants will have received their last dose of study drug in the pivotal study on the day prior to the Week 24/Baseline Visit and were to receive their first dose of study drug for this extension study in the clinic after the participant was determined to be eligible for this extension study and provided informed consent to participate. The administration of the first dose of study drug for MVT-601-3003 was to define enrollment into this study. Study participants were to then take the open-label study treatment orally once daily for 28 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Completed 24 weeks of study drug treatment and study participation in either pivotal study, MVT-601-3001 or MVT-601-3002

Key Exclusion Criteria:

1. Has undergone myomectomy, ultrasound-guided laparoscopic radiofrequency ablation, or any other surgical procedure for fibroids, uterine artery embolization, magnetic resonance-guided focused ultrasound for fibroids, or endometrial ablation for abnormal uterine bleeding at any time during the pivotal study (MVT-601-3001 or MVT-601-3002)
2. Met a withdrawal criterion in the pivotal study (MVT-601-3001 or MVT-601-3002).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 477 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myovant Medical Monitor, Study Director — Myovant Sciences
Locations (130):
- United States (87):
  - Andalusia, Andalusia, Alabama
  - Birmingham, Birmingham, Alabama
  - Mobile, Mobile, Alabama
  - Mesa, Mesa, Arizona
  - Tucson, Tucson, Arizona
  - Little Rock, Little Rock, Arkansas
  - Canoga Park, Canoga Park, California
  - Huntington Beach, Huntington Beach, California
  - La Mesa, La Mesa, California
  - Long Beach, Long Beach, California
  - Los Angeles, Los Angeles, California
  - Norwalk, Norwalk, California
  - Panorama, Panorama City, California
  - San Diego, San Diego, California
  - Denver, Denver, Colorado
  - Lakewood, Lakewood, Colorado
  - Washington, Washington D.C., District of Columbia
  - Aventura, Aventura, Florida
  - Clearwater, Clearwater, Florida
  - DeLand, DeLand, Florida
  - Ft. Lauderdale, Fort Lauderdale, Florida
  - Fort Myers, Fort Myers, Florida
  - Hialeah, Hialeah, Florida
  - Jacksonville, Jacksonville, Florida
  - Jupiter, Jupiter, Florida
  - Loxahatchee, Loxahatchee Groves, Florida
  - Margate, Margate, Florida
  - Miami, Miami, Florida
  - New Port Richey, New Port Richey, Florida
  - Orlando, Orlando, Florida
  - Oviedo, Oviedo, Florida
  - Palm Harbor, Palm Harbor, Florida
  - Saint Cloud, Saint Cloud, Florida
  - Sarasota, Sarasota, Florida
  - Tampa, Tampa, Florida
  - West Palm Beach, West Palm Beach, Florida
  - Weston, Weston, Florida
  - Atlanta, Atlanta, Georgia
  - Augusta, Augusta, Georgia
  - College Park, College Park, Georgia
  - Decatur, Decatur, Georgia
  - Duluth, Duluth, Georgia
  - Norcross, Norcross, Georgia
  - Savannah, Savannah, Georgia
  - Chicago, Chicago, Illinois
  - Naperville, Naperville, Illinois
  - Oakbrook, Oakbrook Terrace, Illinois
  - Shawnee, Shawnee Mission, Kansas
  - Covington, Covington, Louisiana
  - Marrero, Marrero, Louisiana
  - Metairie, Metairie, Louisiana
  - Baltimore, Baltimore, Maryland
  - Towson, Towson, Maryland
  - Canton, Canton, Michigan
  - Detroit, Detroit, Michigan
  - Saginaw, Saginaw, Michigan
  - Lincoln, Lincoln, Nebraska
  - Las Vegas, Las Vegas, Nevada
  - Lawrenceville, Lawrenceville, New Jersey
  - Albuquerque, Albuquerque, New Mexico
  - Brooklyn, Brooklyn, New York
  - New York, New York, New York
  - Williamsville, Williamsville, New York
  - Durham, Durham, North Carolina
  - Raleigh, Raleigh, North Carolina
  - Winston-Salem, Winston-Salem, North Carolina
  - Cincinnati, Cincinnati, Ohio
  - Columbus, Columbus, Ohio
  - Englewood, Englewood, Ohio
  - Philadelphia, Philadelphia, Pennsylvania
  - Bluffton, Bluffton, South Carolina
  - Charleston, Charleston, South Carolina
  - Columbia, Columbia, South Carolina
  - Chattanooga, Chattanooga, Tennessee
  - Memphis, Memphis, Tennessee
  - Beaumont, Beaumont, Texas
  - Dallas, Dallas, Texas
  - Fort Worth, Fort Worth, Texas
  - Houston, Houston, Texas
  - Longview, Longview, Texas
  - San Antonio, San Antonio, Texas
  - Sugar Land, Sugar Land, Texas
  - Webster, Webster, Texas
  - Salt Lake City, Salt Lake City, Utah
  - Norfolk, Norfolk, Virginia
  - Richmond, Richmond, Virginia
  - Spokane, Spokane, Washington
- Belgium (4):
  - La Louvière, La Louvière, Hainaut
  - Gent, Ghent, Oost-vlaanderen
  - Brussels, Brussels
  - Jette, Jette
- Brazil (6):
  - Santo Andre, Santo André, Santo Andre
  - Santo André, Santo André, São Paulo
  - São Bernardo Do Campo, São Bernardo do Campo, São Paulo
  - Sao Paulo, São Paulo, São Paulo
  - Botucatu, Botucatu
  - Porto Alegre, Porto Alegre
- Chile (4):
  - Providencia, Providencia
  - San Ramon, San Ramón
  - Region Metropolitana, Santiago
  - Santiago, Santiago
- Czechia (4):
  - Ceské Budejovice, České Budějovice
  - Jihlava, Jihlava
  - Olomouc, Olomouc
  - Pisek, Písek
- Hungary (6):
  - Gyula, Gyula, Bekes County
  - Kecskemét, Kecskemét, Bács-Kiskun county
  - Debrecen, Debrecen, Hajdú-Bihar
  - Nyíregyháza, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Debrecen, Debrecen
  - Szentes, Szentes
- Italy (5):
  - Catanzaro, Catanzaro
  - Firenze, Florence
  - Roma, Roma
  - Siena, Siena
  - Torino, Torino
- Poland (8):
  - Poznan, Poznan, Greater Poland Voivodeship
  - Skórzewo, Skórzewo, Greater Poland Voivodeship
  - Lublin, Lublin, Lublin Voivodeship
  - Warszawa, Warsaw, Masovian Voivodeship
  - Katowice, Katowice, Silesian Voivodeship
  - Szczecin, Szczecin, West Pomeranian Voivodeship
  - Bialystok, Bialystok
  - Lódz, Lódz, Łódź Voivodeship
- South Africa (6):
  - Centurion, Centurion, Gauteng
  - Roodepoort, Roodepoort, Gauteng
  - Durban, Durban, KwaZulu-Natal
  - Bloemfontein, Bloemfontein
  - Cape Town, Cape Town
  - Port Elizabeth, Port Elizabeth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stewart EA, Al-Hendy A, Lukes AS, Madueke-Laveaux OS, Zhu E, Proehl S, Schulmann T, Marsh EE. Relugolix combination therapy in Black/African American women with symptomatic uterine fibroids: LIBERTY Long-Term Extension study. Am J Obstet Gynecol. 2024 Feb;230(2):237.e1-237.e11. doi: 10.1016/j.ajog.2023.10.030. Epub 2023 Oct 18. PMID 37863160
- [Derived] Al-Hendy A, Lukes AS, Venturella R, Villarroel C, McKain L, Li Y, Wagman RB, Stewart EA. A plain language summary of the long-term relugolix combination therapy study for uterine fibroids. J Comp Eff Res. 2023 Aug;12(8):e230069. doi: 10.57264/cer-2023-0069. Epub 2023 Jul 21. PMID 37477173
- [Derived] Al-Hendy A, Lukes AS, Poindexter AN 3rd, Venturella R, Villarroel C, McKain L, Li Y, Wagman RB, Stewart EA. Long-term Relugolix Combination Therapy for Symptomatic Uterine Leiomyomas. Obstet Gynecol. 2022 Dec 1;140(6):920-930. doi: 10.1097/AOG.0000000000004988. Epub 2022 Nov 2. PMID 36357960

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants who completed their participation in one of the pivotal studies (MVT-601-3001 or MVT-601-3002) were eligible to enroll in this study.
Pre-assignment Details: The study results were presented by treatment group in the pivotal study but all the participants received relugolix plus Estradiol (E2)/Norethindrone Acetate (NETA) in open-label extension study.
Groups:
- Relugolix Plus E2/NETA (Group A): Relugolix 40 mg once daily co-administered with E2 (1 mg) and NETA (0.5 mg) for 24 weeks in the pivotal study followed by 28 weeks of relugolix 40 mg once daily co-administered with E2 (1 mg) and NETA (0.5 mg) in this study.
- Relugolix Plus Delayed E2/NETA (Group B): Relugolix 40 mg monotherapy (once daily) for 12 weeks followed by relugolix 40 mg once daily co-administered with E2 (1mg) and NETA (0.5 mg) for 12 weeks in the pivotal study followed by 28 weeks of relugolix 40 mg once daily co-administered with E2 (1 mg) and NETA (0.5 mg) in this study.
- Placebo (Group C): Relugolix placebo co-administered with E2/NETA placebo for up to 24 weeks in the pivotal study followed by 28 weeks of relugolix 40 mg once daily co-administered with E2 (1 mg) and NETA (0.5 mg) in this study.
Period: Overall Study
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Started | 163 | 150 | 164
Received at Least 1 Dose of Study Drug | 163 | 149 | 164
Completed | 133 | 108 | 122
Not Completed | 30 | 42 | 42
Not completed — Adverse Event | 5 | 5 | 9
Not completed — Protocol deviation | 2 | 1 | 2
Not completed — Lost to Follow-up | 7 | 10 | 10
Not completed — Withdrawal by Subject | 9 | 12 | 11
Not completed — Lack of Efficacy | 2 | 7 | 5
Not completed — Other | 5 | 6 | 5
Not completed — Participants who did not receive any study drug | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Extension Safety Population: all enrolled participants who received any amount of open-label study drug in the open-label extension study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C) | Total
Number analyzed (Participants) | 163 | 149 | 164 | 476
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (5.08) | 42.1 (5.58) | 41.9 (5.43) | 42.2 (5.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 149 | 164 | 476
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 34 | 36 | 108
  Not Hispanic or Latino | 122 | 113 | 126 | 361
  Unknown or Not Reported | 3 | 2 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 7 | 1 | 10
  Asian | 0 | 3 | 0 | 3
  Black or African American | 69 | 81 | 88 | 238
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 85 | 51 | 71 | 207
  Other | 2 | 3 | 2 | 7
  Multiple | 2 | 2 | 1 | 5
  Not Reported | 3 | 2 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 113 | 104 | 117 | 335
  Belgium | 0 | 3 | 1 | 4
  Brazil | 4 | 6 | 2 | 12
  Chile | 5 | 6 | 8 | 19
  Czechia | 4 | 2 | 2 | 8
  Hungary | 6 | 4 | 7 | 17
  Italy | 7 | 5 | 3 | 15
  Poland | 14 | 14 | 19 | 47
  South Africa | 10 | 5 | 5 | 20
Mean Menstrual Blood Loss (MBL) volume [Mean (Standard Deviation); unit: mL] | 248.71 (196.694) | 238.78 (155.332) | 216.01 (123.786) | 234.33 (161.753)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.384 (7.0470) | 30.997 (6.4000) | 32.577 (7.4556) | 31.675 (7.0162)
Bone Mineral Density (BMD) [Mean (Standard Deviation); unit: g/cm^2]
  Lumbar Spine (L1-L4) | 1.186 (0.1599) | 1.225 (0.1730) | 1.239 (0.1573) | 1.217 (0.1645)
  Total Hip | 1.044 (0.1382) | 1.062 (0.1463) | 1.069 (0.1401) | 1.058 (0.1415)
  Femoral Neck | 0.960 (0.1572) | 0.994 (0.1657) | 0.994 (0.1648) | 0.982 (0.1630)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Participants Who Achieved Or Maintained An MBL Volume Of <80 Milliliters (mL) And At Least A 50% Reduction From Baseline MBL Volume At Week 52/End Of Treatment
Description: A responder was a participant who had MBL volume of < 80 mL and at least a 50% reduction from baseline MBL volume over the last 35 days of treatment (up to Week 52). All returned feminine products collected at each clinical visit were analyzed by the alkaline hematin method to obtain the MBL volume. MBL volume was measured over the Week 52/early termination feminine product collection interval (up to 35 days prior to the last dose of treatment). The percentage of participants who were responders are presented.
Time Frame: Week 52/End of Treatment
Population: Extension Study Population: all participants who enrolled and received any amount of open-label study drug in the open-label extension study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 163 | 149 | 164
percentage of participants | 86.50 [80.28 to 91.34] | 79.87 [72.52 to 85.98] | 75.00 [67.65 to 81.42]

2. Secondary Outcome: Change From Pivotal Study Baseline In MBL Volume At Week 52
Description: MBL volume was measured using the alkaline hematin method, which involves chemically measuring the blood content of used feminine products. The volume of MBL is measured in mL and a blood loss of 80 mL or more per cycle is considered diagnostic of heavy menstrual bleeding. The least squares (LS) mean was derived for each treatment group using a mixed-effects model with repeated measure with visit, region, and Baseline MBL as fixed effects.
Time Frame: Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 120 | 103 | 113
mL | -251.6 (16.38) | -219.1 (13.91) | -204.7 (13.31)

3. Secondary Outcome: Percentage Of Participants Who Achieved Or Maintained Amenorrhea Over The Last 35 Days Of Treatment
Description: Amenorrhea was defined as meeting 1 of the following criteria for 2 consecutive visits:
  * No feminine product returned due to reported amenorrhea;
  * No feminine product returned due to reports of spotting/negligible bleeding coupled with other data (participant's paper diary) indicating infrequent non-cyclic bleeding/spotting; and
  * Feminine product collection with a negligible observed MBL volume coupled with data (participant's paper diary) indicating infrequent non-cyclic bleeding/spotting.
Time Frame: Week 24 up to last 35 days of treatment (up to Week 52)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 163 | 149 | 164
percentage of participants | 70.55 [62.92 to 77.42] | 68.46 [60.35 to 75.82] | 57.93 [49.98 to 65.58]

4. Secondary Outcome: Percentage Of Participants With A Hemoglobin Level ≤10.5 Gram/Deciliter (g/dL) At Pivotal Study Baseline Who Achieved An Increase Of >2 g/dL From Pivotal Study Baseline At Week 52
Description: Blood samples were collected from participants for hemoglobin measurements. Percentages are based on number of participants with hemoglobin ≤10.5 g/dL at pivotal study Baseline and reported at Week 52.
Time Frame: Week 52
Population: Extension Study Population with a hemoglobin level ≤10.5 g/dL at pivotal study baseline: all participants who enrolled and received any amount of open-label study drug in the open-label extension study and who had a hemoglobin level ≤10.5 g/dL at pivotal study baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 39 | 38 | 38
percentage of participants | 58.97 [42.10 to 74.43] | 78.95 [62.68 to 90.45] | 42.11 [26.31 to 59.18]

5. Secondary Outcome: Number Of Participants With Hemoglobin Increase Of ≥1 g/dL From Pivotal Study Baseline At Week 52 Among Those With A Hemoglobin Concentration Below Lower Limit Of Normal At Pivotal Baseline
Description: Blood samples were collected from participants for hemoglobin measurements. Percentages are based on number of participants with hemoglobin concentration below the lower limit of normal (11.6 g/dL) at pivotal study Baseline and reported at Week 52.
Time Frame: Week 52
Population: Extension Study Population with a hemoglobin level below lower limit of normal at pivotal study baseline: all participants who enrolled and received any amount of open-label study drug in the open-label extension study and who had a hemoglobin level below lower limit of normal at pivotal study baseline.
Measure: Number; unit: participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 89 | 96 | 98
participants | 56 | 60 | 45

6. Secondary Outcome: Change From Pivotal Study Baseline In Hemoglobin Concentration At Week 52
Description: Blood samples were collected from participants for hemoglobin measurements. The LS mean was derived for each treatment group using a mixed-effects model with repeated measure.
Time Frame: Week 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 39 | 38 | 38
g/dL | 2.7 (0.24) | 3.0 (0.23) | 1.9 (0.22)

7. Secondary Outcome: Change From Pivotal Study Baseline In The UFS-QoL Symptom Severity Scale At Week 52
Description: Transformed score ranges from 0 to 100 based on Likert scale (none of time, a little of time, some of the time, most of the time, and all of the time). Lower score indicates less distress and higher score indicates greater distress. A negative change from baseline indicates improvement. The LS mean was derived for each treatment group using a mixed-effects model with repeated measure.
Time Frame: Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 129 | 108 | 120
score on a scale | -37.3 (2.47) | -38.2 (2.77) | -35.0 (2.48)

8. Secondary Outcome: Change From Pivotal Study Baseline In The UFS-QoL Score Health-Related Quality of Life Subscales Score At Week 52
Description: Assessed using the UFS-QoL questionnaire. The UFS-QoL subscale scores include items related to uterine fibroid-associated limitations/impairment in activities, revised activities, concern, energy/mood, control, self-consciousness, and sexual function. The scores were transformed to normalized scores. Transformed score ranges from 0 to 100. Higher scores are indicative of better health-related quality of life (high = good). The LS mean was derived for each treatment group using a mixed-effects model with repeated measure.
Time Frame: Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 129 | 108 | 120
score on a scale
  Concern | 56.4 (2.92) | 56.4 (3.10) | 51.2 (3.10)
  Activities | 47.8 (2.72) | 46.9 (2.82) | 45.2 (2.81)
  Revised activities | 49.2 (2.78) | 48.0 (2.97) | 46.9 (2.85)
  Energy/mood | 35.6 (2.67) | 38.6 (2.88) | 36.5 (2.79)
  Control | 33.0 (2.69) | 36.4 (2.82) | 32.2 (2.91)
  Self-conscious | 31.2 (3.06) | 35.4 (3.40) | 31.0 (3.14)
  Sexual function | 22.7 (3.40) | 22.0 (3.87) | 24.1 (3.62)

9. Secondary Outcome: Change From Pivotal Study Baseline In The UFS-QoL Score By Health-Related Quality of Life Total Score At Week 52
Description: Assessed using the UFS-QoL Questionnaire. The UFS-QoL total score was the sum of the subscales (concern, activities, revised activities, energy/mood, control, self-conscious, and sexual function). The raw scores were transformed to normalized scores. Transformed score ranges from 0 to 100. Higher scores are indicative of better health-related quality of life (high = good). The LS mean was derived for each treatment group using a mixed-effects model with repeated measure.
Time Frame: Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 129 | 108 | 120
score on a scale | 40.4 (2.50) | 41.7 (2.68) | 39.0 (2.63)

10. Secondary Outcome: Change From Pivotal Study Baseline In The Uterine Fibroid Symptom Health-Related Quality of Life (UFS-QoL) Bleeding And Pelvic Discomfort (BPD) Scale At Week 52
Description: The BPD scale has been derived from the UFS-QoL symptom severity scale. The scale consists of the following 3 symptoms proximal to uterine fibroids that are experienced by most participants: heavy bleeding during the menstrual period (Question 1), passing blood clots during the menstrual period (Question 2), and feeling tightness or pressure in the pelvic area (Question 5). Raw scores were transformed to a normalized score, with a range of possible scores from 0 to 100 (none of time, a little of time, some of the time, most of the time, and all of the time), where higher scores values are indicative of greater distress and lower scores are indicative of minimal distress. The LS mean was derived for each treatment group using a mixed-effects model with repeated measure.
Time Frame: Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 129 | 108 | 120
score on a scale | -51.3 (2.66) | -51.6 (3.11) | -48.6 (2.76)

11. Secondary Outcome: Change From Pivotal Study Baseline In Uterine Volume At Week 52
Description: Volume of the uterus was measured by transvaginal or transabdominal ultrasound. The LS mean was derived for each treatment group using a mixed-effects model with repeated measure.
Time Frame: Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm^3
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 136 | 110 | 119
cm^3 | -73.31 (14.471) | -91.67 (20.143) | -37.62 (14.541)

12. Secondary Outcome: Change From Pivotal Study Baseline In Uterine Fibroid Volume At Week 52
Description: Volume of the primary uterine fibroid was measured by transvaginal or transabdominal ultrasound. The LS mean was derived for each treatment group using a mixed-effects model with repeated measure.
Time Frame: Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm^3
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 131 | 103 | 117
cm^3 | -31.84 (5.353) | -28.18 (5.523) | -17.07 (5.726)

13. Secondary Outcome: Percent Change From Pivotal Study Baseline In Bone Mineral Density (BMD) At The Lumbar Spine (L1-L4), Femoral Neck, And Total Hip At Week 52
Description: Assessed by dual-energy X-ray absorptiometry (DXA) scan at the lumbar spine (L1-L4), total hip, and femoral neck at pivotal study Baseline and at Week 52. The scans were read by the central radiology laboratory in accordance with the imaging charter. The same DXA machine was used at the local imaging center at each site and operated in the same scan mode for all images procured for an individual participant. All images were submitted for central reading. The central radiology laboratory collected and evaluated all DXA scans for acceptability and measured BMD. The LS mean was derived for each treatment group using a mixed-effects model with repeated measure.
Time Frame: Week 52
Population: Extension Safety Population: all enrolled participants who received any amount of open-label study drug in the open-label extension study. The overall number of participants analyzed is then umber of patients at baseline. The number analyzed at each location is the number of patients included in summary statistics for that location and timepoint.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 163 | 149 | 164
percentage change
  Lumbar Spine (L1-L4): number analyzed (Participants) | 132 | 108 | 120
  Lumbar Spine (L1-L4) | -0.804 (0.2803) | -2.045 (0.2679) | -0.775 (0.2781)
  Total Hip: number analyzed (Participants) | 129 | 105 | 121
  Total Hip | -0.153 (0.2337) | -0.842 (0.2308) | -0.065 (0.2086)
  Femoral Neck: number analyzed (Participants) | 129 | 105 | 121
  Femoral Neck | -0.575 (0.3208) | -0.513 (0.4503) | 0.004 (0.3886)

14. Secondary Outcome: Change From Pivotal Study Baseline In Predose Serum E2 Concentrations At Week 52
Description: Blood samples were collected from participants at predose for E2 measurements. These were analyzed at a central laboratory.
Time Frame: Week 52
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 135 | 114 | 125
pg/mL | -21.83 (91.525) | -33.77 (106.407) | -29.99 (81.465)

15. Other Pre Specified Outcome: Change From Pivotal Study Baseline In European Quality Of Life Five Dimension Five Level (EQ-5D-5L) Scale At Week 52
Description: The EQ-5D-5L scale is a standardized instrument for use as a measure of health outcomes. Mobility, self-care, usual activities, pain/discomfort, and anxiety/depression were each assessed on 5-point categorical scales of no problems to unable to complete specified activity, or no pain/discomfort to extreme pain/discomfort, or not anxious/depressed to extremely anxious/depressed. The change from baseline is summarized by amount of improvement (1-4 categories), amount of deterioration (1-4 categories), or no change.
Time Frame: Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 127 | 108 | 117
Participants
  Mobility - 4 Category deterioration | 0 | 0 | 0
  Mobility - 3 Category deterioration | 0 | 1 | 0
  Mobility - 2 Category deterioration | 2 | 0 | 0
  Mobility - 1 Category deterioration | 3 | 5 | 4
  Mobility - No change | 102 | 89 | 99
  Mobility - 1 Category improvement | 15 | 9 | 10
  Mobility - 2 Category improvement | 5 | 3 | 4
  Mobility - 3 Category improvement | 0 | 1 | 0
  Mobility - 4 Category improvement | 0 | 0 | 0
  Self-care - 4 Category deterioration | 0 | 0 | 0
  Self-care - 3 Category deterioration | 0 | 0 | 0
  Self-care - 2 Category deterioration | 0 | 1 | 0
  Self-care - 1 Category deterioration | 1 | 1 | 2
  Self-care - No change | 122 | 105 | 108
  Self care - 1 Category improvement | 3 | 0 | 5
  Self care - 2 Category improvement | 1 | 1 | 1
  Self care - 3 Category improvement | 0 | 0 | 0
  Self care - 4 Category improvement | 0 | 0 | 1
  Usual activities - 4 Category deterioration | 0 | 0 | 0
  Usual activities - 3 Category deterioration | 0 | 1 | 0
  Usual activities - 2 Category deterioration | 3 | 0 | 2
  Usual activities - 1 Category deterioration | 4 | 2 | 4
  Usual activities - No change | 91 | 71 | 73
  Usual activities - 1 Category improvement | 15 | 22 | 22
  Usual activities - 2 Category improvement | 10 | 10 | 12
  Usual activities - 3 Category improvement | 3 | 2 | 3
  Usual activities - 4 Category improvement | 1 | 0 | 1
  Pain/discomfort - 4 Category deterioration | 0 | 0 | 0
  Pain/discomfort - 3 Category deterioration | 0 | 1 | 2
  Pain/discomfort - 2 Category deterioration | 3 | 2 | 0
  Pain/discomfort - 1 Category deterioration | 17 | 8 | 10
  Pain/discomfort - No change | 46 | 45 | 45
  Pain/discomfort - 1 Category improvement | 37 | 31 | 37
  Pain/discomfort - 2 Category improvement | 16 | 14 | 17
  Pain/discomfort - 3 Category improvement | 8 | 6 | 6
  Pain/discomfort - 4 Category improvement | 0 | 1 | 0
  Anxiety/depression - 4 Category deterioration | 0 | 0 | 1
  Anxiety/depression - 3 Category deterioration | 0 | 0 | 0
  Anxiety/depression - 2 Category deterioration | 4 | 3 | 5
  Anxiety/depression - 1 Category deterioration | 11 | 20 | 12
  Anxiety/depression - No change | 79 | 53 | 69
  Anxiety/depression - 1 Category improvement | 24 | 25 | 17
  Anxiety/depression - 2 Category improvement | 8 | 7 | 11
  Anxiety/depression - 3 Category improvement | 0 | 0 | 1
  Anxiety/depression - 4 Category improvement | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Week 24 up to Week 52
Description: Extension Safety Population: all enrolled participants who received any amount of open-label study drug in the open-label extension study.
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/149 | 0/164
Serious Adverse Events (participants affected / at risk) | 1/163 | 5/149 | 11/164
Other Adverse Events (participants affected / at risk) | 22/163 | 12/149 | 38/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relugolix Plus E2/NETA (Group A) (N=163) | Relugolix Plus Delayed E2/NETA (Group B) (N=149) | Placebo (Group C) (N=164)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 2
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Relugolix Plus E2/NETA (Group A) (N=163) | Relugolix Plus Delayed E2/NETA (Group B) (N=149) | Placebo (Group C) (N=164)
Headache (Nervous system disorders) | 6 | 7 | 11
Hot flush (Vascular disorders) | 4 | 0 | 13
Nasopharyngitis (Infections and infestations) | 10 | 3 | 8
Hypertension (Vascular disorders) | 2 | 3 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT03412890/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/90/NCT03412890/SAP_001.pdf